CLINICAL TRIAL: NCT01186315
Title: Developing a Computer-Based Intervention to Enhance Behavioral Treatments for PTSD and Addiction
Brief Title: Post-traumatic Stress Disorder (PTSD), Addiction, and Virtual Reality
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Duke University (Other)
Collaborators: United States Department of Defense (U.S. Federal Agency); Telemedicine & Advanced Technology Research Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Pro00011730; 01445 (Other: Durham VAMC Institutional Review Board); 08144019 (Other Grant/Funding Number: US Department of Defense)
Record Dates: First submitted 2010-08-19; First posted 2010-08-23 (Estimated); Last update posted 2014-08-21 (Estimated); Status verified 2014-08

CONDITIONS: Substance Use Disorders; Posttraumatic Stress Disorder
Keywords: Addiction; Posttraumatic Stress; substance abuse and posttraumatic stress
MeSH Terms: conditions — Substance-Related Disorders; Stress Disorders, Post-Traumatic; Behavior, Addictive | interventions — Implosive Therapy

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Prolonged Exposure therapy (Active Comparator): These treatments include repeated exposure to intrusive trauma-related memories in a safe and structured manner designed to reduce emotional arousal and facilitate processing of trauma-related memories.
  Interventions: Behavioral: Prolonged Exposure Therapy
- Exposure therapy + VR/ER (Experimental): prolonged exposure therapy plus virtual reality (VR) based cue exposure/extinction software and cellular phone-based computerized extinction reminder (CER) technology for use in high-risk situations outside treatment sessions.
  Interventions: Behavioral: Prolonged Exposure therapy + VR/ER

INTERVENTIONS:
Behavioral: Prolonged Exposure Therapy — These treatments include repeated exposure to intrusive trauma-related memories in a safe and structured manner designed to reduce emotional arousal and facilitate processing of trauma-related memories.
  Other Names: Exposure Therapy
  Arms: Prolonged Exposure therapy
Behavioral: Prolonged Exposure therapy + VR/ER — The therapy includes repeated exposure to intrusive trauma-related memories in a safe and structured manner designed to reduce emotional arousal and facilitate processing of trauma-related memories and adding in virtual reality (VR)-based exposure to cues for marijuana, cocaine, heroin, cigarette, and/or alcohol use & CER used outside treatment sessions in response to VR exposure (available 24 hours per day/7 days per week) to high-risk contexts for drug use
  Other Names: virtual reality; exposure therapy; CER; VR; cell-phone based computerized extinction reminder
  Arms: Exposure therapy + VR/ER

SUMMARY:
Eligible veterans, National Guardsmen & Reservists with post-traumatic stress disorder (PTSD) and problems with addiction will be randomly assigned to one of two treatment conditions. All participants will undergo exposure therapy, a gold standard behavioral treatment for PTSD for 10 weeks. In addition to exposure therapy, some participants will be randomly assigned to receive (1) virtual reality (VR)-based exposure to cues for marijuana, cocaine, heroin, cigarette, and/or alcohol use, and (2) cellular phone-based reminders of learning (extinction reminders, or, ERs) to VR exposure (available 24 hours per day/7 days per week) to high-risk contexts for drug use. The main hypothesis is that those participants who receive exposure therapy + VR/ERs will demonstrate less substance use and lower PTSD symptoms during treatment, at post-treatment, and at follow-up than those participants who only receive exposure therapy. At study completion, a total of 123 subjects signed consent.

DETAILED DESCRIPTION:
Veterans, National Guardsmen, & Reservists with post-traumatic stress disorder (PTSD) and problems with addiction need a wider array of treatment options than what is currently available. The present project offers the promise of a complementary approach that uses computer-based interventions to augment exposure therapy for veterans with both PTSD and use alcohol, nicotine and/or other substances. If this new intervention is found to be efficacious in the present project, it would provide an alternative to standard treatment for a growing number of veterans who are at risk for lifetime problems with PTSD and addiction, but who may be unwilling to begin usual psychotherapy. This direct way of training new behavior in the clinic and extending learning into the real world is missing in treatments for many medical and psychiatric conditions. As such, the impact of this project could extend into treatment of a wide variety of other chronic conditions for which more powerful new treatments are needed. Veterans will be recruited from the Durham Veterans Affairs Medical Center (Durham VAMC) and local community.

Participants (N = 60) meeting full criteria for current diagnoses of both PTSD and at least one SUD were to be recruited through the Durham Veterans Affairs Medical Center (Durham VAMC). 100 participants were to be enrolled (sign the consent form) in order to identify 60 who meet inclusion/exclusion criteria. Actually 123 subjects signed consent and 38 subjects are considered ITT (intent to treat-met inclusion/exclusion criteria, randomized and showed to their first therapy session). Participants were randomly assigned to one of two treatment conditions-exposure therapy alone or exposure therapy + virtual reality (VR)-based exposure to cues for marijuana, cocaine, heroin, cigarette, and/or alcohol use, and (2) cellular phone-based reminders of learning (extinction reminders, or, ERs) to VR exposure. Matching between treatment groups was based on age, gender, severity of PTSD and substance use. In addition, to control for differential dropout and other changes in treatment due to cell phone use in the VR/ER condition, participants in the control condition also carried cell phones, and were randomly called three times a day via the automated server (same as the VR/ER condition). These calls were completed for assessment only, to obtain real time self-reports of substance use and cravings (without the ER). Comprehensive assessments were conducted at pre-treatment, 10 weeks (post-treatment), and at a 6-month follow-up.

The goals of this project are to examine the acceptability and feasibility of the complementary treatment and evaluate the effects of the complementary intervention on PTSD and substance use.

ELIGIBILITY:
Inclusion Criteria:

* Meets SCID-I criteria for PTSD; criterion A stressor must be deployment related, and substance dependence; primary substance of dependence is cocaine, heroin, alcohol, cigarettes, or marijuana
* Must be a Veteran
* Consents to outpatient treatment for PTSD and drug addiction

Exclusion Criteria:

* Full criteria met for current manic episode or psychotic disorder through using SCID-I interviews
* Pregnant at time of treatment
* IQ less than 70; unable to give consent; can not read
* current and chronic absence of shelter
* impending jail/prison for more than three weeks
* Court order to treatment, court order to treatment or to jail, or agency order to treatment or loss of child custody (due to inability to freely drop-out of treatment)
* Refuses to discontinue current mental health or drug abuse behavioral treatment (i.e., psychotherapy) or random assignment
* Suicide attempt or self-harm in the past 6 months

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 38 (Actual)
Dates: Start 2008-12; Primary Completion 2013-10 (Actual); Study Completion 2013-12 (Actual)

PRIMARY OUTCOMES:
Acceptability/feasibility (e.g., retention) of the novel intervention | 10 weeks + 6 month follow-up
  Acceptability/feasibility of exposure therapy + VR/ER will be evidenced by rates of session attendance, retention, and exit interview ratings
Change in PTSD symptoms | Pre treatment, 10 weeks, post treatment, 6 month follow-up
  Self-report measures of PTSD symptoms [e.g. The Davidson Trauma Scale (DTS)]and interview measures [e.g. Structured interview for DSM-IV, Axis I (SCID-I), Clinician Administered PTSD Scale (CAPS)]
Change in substance use | Pre Treatment, Post 10 Week Treatment, and 6 month Follow Up
  Self report measures of substance use: (e.g. Fagerström Test for Nicotine Dependence, Smoking Effects Questionnaire, Alcohol Craving Questionnaire, Heroin Craving Questionnaire, Cocaine Craving Questionnaire) and Interview Measures: [e.g. Structured Clinical Interview for DSM-IV, Axis I (SCID-I); Addiction Severity Index (ASI); Time Line Follow-back Assessment Method]

SECONDARY OUTCOMES:
Biochemical measures | Pre Treatment, Post Treatment, Follow Up, During 10 weeks of Treatment
  * Urinalysis testing is done using the Biosite Diagnostics Triage Meter Plus within 24 hours for cocaine, marijuana, opiates, amphetamines, and benzodiazepines. Will be thrice weekly during 10 weeks of treatment.
  * Breathalyzer is done Pre Treatment, Post Treatment, Follow Up and before sessions during treatment.

CONTACTS AND LOCATIONS:
Overall Officials: Zachary Rosenthal, PhD, Principal Investigator — Duke University
Locations (1):
- Duke University Medical Center, Durham, North Carolina, United States

REFERENCES:
- [Background] Hoge CW, Castro CA, Messer SC, McGurk D, Cotting DI, Koffman RL. Combat duty in Iraq and Afghanistan, mental health problems, and barriers to care. N Engl J Med. 2004 Jul 1;351(1):13-22. doi: 10.1056/NEJMoa040603. PMID 15229303
- [Background] Najavits LM, Weiss RD, Shaw SR, Muenz LR. "Seeking safety": outcome of a new cognitive-behavioral psychotherapy for women with posttraumatic stress disorder and substance dependence. J Trauma Stress. 1998 Jul;11(3):437-56. doi: 10.1023/A:1024496427434. PMID 9690186
- [Background] McLellan AT, Luborsky L, Woody GE, O'Brien CP. An improved diagnostic evaluation instrument for substance abuse patients. The Addiction Severity Index. J Nerv Ment Dis. 1980 Jan;168(1):26-33. doi: 10.1097/00005053-198001000-00006. PMID 7351540
- [Background] Seal KH, Bertenthal D, Miner CR, Sen S, Marmar C. Bringing the war back home: mental health disorders among 103,788 US veterans returning from Iraq and Afghanistan seen at Department of Veterans Affairs facilities. Arch Intern Med. 2007 Mar 12;167(5):476-82. doi: 10.1001/archinte.167.5.476. PMID 17353495
- [Result] Zlotnick C, Najavits LM, Rohsenow DJ, Johnson DM. A cognitive-behavioral treatment for incarcerated women with substance abuse disorder and posttraumatic stress disorder: findings from a pilot study. J Subst Abuse Treat. 2003 Sep;25(2):99-105. doi: 10.1016/s0740-5472(03)00106-5. PMID 14629992
- [Result] Koenen KC, Hitsman B, Lyons MJ, Stroud L, Niaura R, McCaffery J, Goldberg J, Eisen SA, True W, Tsuang M. Posttraumatic stress disorder and late-onset smoking in the Vietnam era twin registry. J Consult Clin Psychol. 2006 Feb;74(1):186-90. doi: 10.1037/0022-006X.74.1.186. PMID 16551156